CLINICAL TRIAL: NCT03445078
Title: Correction of Selenium Deficiency Has Effect on Thyroid Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liuyanping, nutrition physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Liuyanping4
Record Dates: First submitted 2018-02-07; First posted 2018-02-26 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Selenium Deficiency

STUDY DESIGN:
Intervention Model Description: 20 participants with selenium deficiency (confirmed in previous phase (ID: Liuyanping3)) will be recruited to receive selenium-rich corn powder (20g/d, offering selenium 100μg/d) and ordinary corn powder (20g/d, offering selenium < 0.5μg/d ) in two different sequences (10 subjects each) with a four-week washout period.Plasma samples were obtained at different time points before and after administration of the selenium-rich corn powder and ordinary corn powder.
Who Masked: Participant
Masking Description: All participants will be blinded. Both the selenium-rich corn powder and the ordinary corn powder (placebo) have the same smell, color and taste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): Participants will be administered firstly selenium-rich corn powder 20g/d for 1 month and ordinary corn powder 20g/d for another month subsequently with a month washout period.
  Interventions: Dietary Supplement: selenium supplementation; Dietary Supplement: ordinary corn powder
- B (Placebo Comparator): Participants will be administered firstly ordinary corn powder 20g/d for 1 month and selenium-rich corn powder 20g/d for another month subsequently with a month washout period.
  Interventions: Dietary Supplement: selenium supplementation; Dietary Supplement: ordinary corn powder

INTERVENTIONS:
Dietary Supplement: selenium supplementation — administration of selenium-rich corn powder 20g/d offering selenium 100μg/d
Dietary Supplement: ordinary corn powder — ordinary corn powder,20g/d(selenium contain <0.5ug/20g).
  Other Names: low selenium

SUMMARY:
Previous literature has found potential association between selenium deficiency and inactivated glutathione peroxidase and deiodinase, which may contribute to subsequent elevation of T4 and ratio of T4/T3. Conduction of a case-control study (ID: Liuyanping3) has been applied on Clinicaltrials.gov to further elucidate effect of selenium deficiency on thyroid function. Based on its data, the investigators will perform a randomized, placebo-controlled,single-blinded crossover study on 20 participants with selenium deficiency to verify health consequence of selenium.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of selenium deficiency through serum selenium test in previous phase (ID: Liuyanping3) of the study
* Should have stable body weight in the latest 3 months;
* Should be not prescribed with thyroid hormone replacement therapy
* Should be without medical history of thyroid surgery or iodine radiotherapy
* Should have normal FT3, FT4 and TSH.

Exclusion Criteria:

* Clinical diagnosis of acute critical illness in the latest 1 year
* Have had weight fluctuation by more than 5%
* Eating disorders
* Neuropsychological disorders
* Allergy to corn or yeast

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
comparison of thyroid function | plasma sample will be collected at -1w/4w/8w/12w
  comparison of thyroid function between administration of selenium supplementation and placebo

SECONDARY OUTCOMES:
comparison of serum selenium | plasma sample will be collected at -1w/4w/8w/12w
  comparison of serum selenium between administration of selenium supplementation and placebo
comparison of erythrocyte glutathione peroxidase activity | plasma sample will be collected at -1w/4w/8w/12w
  comparison of erythrocyte glutathione peroxidase activity between administration of selenium supplementation and placebo
comparison of serum deiodinase activity | plasma sample will be collected at -1w/4w/8w/12w
  comparison of serum deiodinase activity between administration of selenium supplementation and placebo